CLINICAL TRIAL: NCT06203314
Title: Prospective Cohort Study on Epstein-Barr Virus Antibody and Cancer Risks
Brief Title: Epstein-Barr Virus and Cancer Risks
Acronym: EBVCR
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Jia wei-hua, Professor, Sun Yat-sen University
Other Study IDs: EBV-PRO-001
Record Dates: First submitted 2023-12-29; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: EBV; Prospective study; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zhongshan cohort, Guangdong, China: 30-59 years old healthy participants in Zhongshan city.
  Interventions: Other: Diagnostic test: EBV antibody tests
- Wuzhou cohort, Guangxi, China: 30-69 years old healthy participants in Wuzhou city.
  Interventions: Other: Diagnostic test: EBV antibody tests

INTERVENTIONS:
Other: Diagnostic test: EBV antibody tests — Participants underwent several EBV antibody tests, including VCA-IgA, EBNA1-IgA, etc.

SUMMARY:
The goal of this prospective cohort study is to investigate the associations between Epstein-Barr Virus (EBV) antibody levels and the risk of overall and site-specific cancer types in Southern China. The main questions it aims to answer are:

Question 1: In addition to the established EBV-associated cancer types, such as lymphomas, nasopharyngeal carcinoma, and stomach cancer, whether EBV is associated with other cancer types? Question 2: What's the cancer burden attributed to EBV in Southern China?

DETAILED DESCRIPTION:
Growing molecular evidence suggests the involvement of EBV in various cancers, however, comprehensive epidemiological evidence is still lacking. In this study, researchers conducted a population-based prospective cohort study to investigate the associations between EBV antibodies and the risk of overall and site-specific cancer types in Southern China. All the participants underwent EBV antibody tests at enrollment and were subsequently followed up annually for cancer incidence, vital status, and immigration status. The primary objective of this study was to provide prospective evidence for the role of EBV in multiple cancers, shedding light on the etiology of a broad range of common EBV-associated cancers.

ELIGIBILITY:
Inclusion Criteria:

* Subject residents in Zhongshan or Wuzhou City;
* Subject has no medical record of prevalent cancer;
* Subject has psychical condition and well consciousness, and willingness to accept and cooperate with the study's follow-up procedures.

Exclusion Criteria:

* Subject has heavy cardiovascular, liver, or kidney disease;
* Subject has prevalent cancer.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30-69 years old healthy residences in Zhongshan City and Wuzhou City.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2008-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer incidence | 10 years
  The primary outcome of the study was the diagnosis of any type of cancer. The cancer type for each participant was defined as their initial and primary cancer diagnosis.

SECONDARY OUTCOMES:
All-cause mortality | 10 years
  The participants were followed up annually for cancer incidence, vital status and immigration status through the Cancer Registry, Death Registry, and Population Registry of local regions.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

IPD SHARING:
Plan to Share IPD: No
In order to prioritize and uphold participant confidentiality and privacy, we have chosen not to provide Individual Participant Data (IPD). Our commitment is to ensure the highest level of protection for the sensitive information of our participants, aligning with ethical principles and privacy regulations. This decision is made to safeguard the well-being and privacy of the individuals involved in the study.